CLINICAL TRIAL: NCT05279820
Title: Full Versus Partial Pulpotomy in the Management of Teeth With Clinical Diagnosis of Irreversible Pulpits: A Randomized Clinical Trial
Brief Title: Comparative Study of the Outcome of Partial and Full Pulpotomy in Irreversible Pulpits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 329/2021
Record Dates: First submitted 2021-11-28; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Carious Exposure of Pulp; Irreversible Pulpitis; Pulpotomy
Keywords: irreversible pulpits; Pulpotomy; Outcome

STUDY DESIGN:
Intervention Model Description: The study will run concurrently and the participants will randomly distributed between the two interventions using a block randomization procedure
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant will not be informed whether the treatment performed was partial or full pulpotomy the outcome assessor will be blinded to the type of treatment performed, and evaluation of the radiographs will include masking the crown so that the procedure cannot be identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial Pulpotomy (Active Comparator): After pulp exposure 2-3 mm of the pulp tissue will be amputated, a calcium silicate based material will be placed over the pulp and the tooth will be restored.
  Interventions: Procedure: Partial pulpotomy
- Full Pulpotomy (Active Comparator): After pulp exposure the entire coronal pulp to the level of canal orifices will be amputated , calcium silicate based material will be placed over the pulp and the tooth will be restored.
  Interventions: Procedure: Full Pulpotomy

INTERVENTIONS:
Procedure: Partial pulpotomy — Partial pulp tissue amputation
  Arms: Partial Pulpotomy
Procedure: Full Pulpotomy — Full Pulpotomy
  Arms: Full Pulpotomy

SUMMARY:
This study aims at comparing the outcome of partial pulpotomy and full pulpotomy in the management of carious pulp exposures in permanent teeth with a clinical diagnosis of irreversible pulpits. The primary outcome is resolution of symptoms and the secondary outcome is clinical and radiographic normality at 1 and 2 years follow up.

The study design will be a double blind randomized clinical trial.

DETAILED DESCRIPTION:
Aim: to compare the outcome of partial and full pulpotomy in managing carious pulp exposures in mature permanent teeth with symptoms of irreversible pulpitis

Methods: Assuming a 10% difference in the success rate in favor of pulpotomy, with 80% power and accounting for possible 10% attrition, the minimum sample size required is estimated to be 80 teeth in 80 patients in every arm.

Patients referred to the postgraduate Endodontic clinic for management of deep carious lesions with symptoms of irreversible pulpits will be assessed for inclusion in the study according to preset inclusion criteria. After a written informed consent baseline demographics of patients and teeth will be recorded.

Pulpotomy (partial or full using block randomization) will be performed under aseptic procedures and the tooth will be permanently restored. Post operative baseline radiographs will be taken.

Primary outcome will be assessed after 48 hours. secondary outcome will be assessed at 6 months, 1 year and 2 years post operatively.

Data of outcome and effect of preoperative and intraoperative variables on the outcome will be compared statistically using appropriate tests

ELIGIBILITY:
Inclusion Criteria:

* Mature permanent tooth
* Deep caries extending more than two thirds of dentine or exposing the pulp
* Tooth responds positively to cold test
* Clinical symptoms of irreversible pulpits
* Tooth is restorable and can be restored with coronal restoration
* Bleeding normally is confirmed after pulp exposure
* hemostasis could be achieved within 8 minutes

Exclusion Criteria:

* Non restorable teeth
* necrotic teeth
* hemostasis could not be achieved within 8 minutes

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Post operative pain level measured by visual analogy scale from 0-10 | 48 hours
  scale from 0-10
Post operative pain level measured by a numerical scale from 0-10 | 48 hours
  scale from 0-10

SECONDARY OUTCOMES:
Clinical success as measured by clinical examination | 6, 12, 24 months
  The tooth should be pain free, no sinus tract or swelling, no tenderness to palpation as determined by clinical examination
Radiographic success as evaluated by periapical x-rays | 6, 12, 24 months
  There should be no evidence of bone resorption or root resorption on the x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Nessrin Taha, PhD, Study Chair — Jordan University of Science and Technology
Locations (1):
- Jordan University of science and technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
Until the time of completion of the study, ankylosis of data and submission for publication, then data can be provided to other researchers

REFERENCES:
- [Background] Taha NA, About I, Sedgley CM, Messer HH. Conservative Management of Mature Permanent Teeth with Carious Pulp Exposure. J Endod. 2020 Sep;46(9S):S33-S41. doi: 10.1016/j.joen.2020.06.025. PMID 32950193